CLINICAL TRIAL: NCT02556463
Title: A Phase I, First-Time-in-Human Study of MEDI9197, a TLR 7/8 Agonist, Administered Intratumorally as a Single Agent in Subjects With Solid Tumors or CTCL and in Combination With Durvalumab and/or Palliative Radiation in Subjects With Solid Tumors
Brief Title: A Study of MEDI9197 in Subjects With Solid Tumors or CTCL and in Combination With Durvalumab and/or Palliative Radiation in Subjects With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company strategy
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6410C00001
Record Dates: First submitted 2015-09-01; First posted 2015-09-22 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Solid Tumors; CTCL; Cancer
Keywords: MEDI9197; TLR 7/8 Agonist; Durvalumab; MEDI4736; Imfinzi
MeSH Terms: conditions — Neoplasms | interventions — MEDI9197; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Escalation MEDI9197 (Experimental): MEDI9197
  Interventions: Drug: MEDI9197
- Escalation MEDI9197 with durvalumab (Experimental): MEDI9197 in combination with durvalumab
  Interventions: Drug: MEDI9197; Biological: durvalumab
- Escalation MEDI9197 durvalumab radiation (Experimental): MEDI9197 in combination with durvalumab and palliative radiation
  Interventions: Drug: MEDI9197; Biological: durvalumab
- MEDI9197 with palliative radiation (Experimental): MEDI9197 in combination with palliative radiation
  Interventions: Drug: MEDI9197

INTERVENTIONS:
Drug: MEDI9197 — Subjects will receive MEDI9197 (every 4 weeks) as monotherapy (or MEDI9197 every 8 weeks + durvalumab every 4 weeks)(PA6)
Biological: durvalumab — Subjects will receive durvalumab every 4 weeks
  Other Names: MEDI4736
  Arms: Escalation MEDI9197 durvalumab radiation; Escalation MEDI9197 with durvalumab

SUMMARY:
To evaluate MEDI9197 when administered by intratumoral injection to subjects with solid tumors and in combination with durvalumab in subjects with solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label study to evaluate the TLR 7/8 agonist MEDI9197 delivered by IT injection to subjects with solid tumors and in combination with durvalumab in subjects with solid tumors. The study has a dose escalation design using mTPI-2 to evaluate a range of doses.

ELIGIBILITY:
Inclusion Criteria for All Subjects (Parts 1, 2 and 3)

1. Written informed consent and any locally required authorizations.
2. Male and female subjects at least 18 years at the time of screening.
3. Adequate organ function within 14 days of enrollment confirmed by laboratory results.
4. Systemic corticosteroids at doses exceeding 12 mg/day prednisone or equivalent.
5. ECOG 0 or 1.
6. Highly effective method of contraception from the date of the screening pregnancy test, and continued precautions for 6 months after the final dose of investigational product.
7. Baseline Child-Pugh Score of A1 to B7.
8. Life expectancy ≥ 12 weeks, as estimated by Royal Marsden Hospital Score of 0 or 1 at baseline.
9. Subjects with hepatocellular carcinoma (HCC) are eligible if the tumor is defined as nodular type 1 or 2 only.

   Additional Inclusion Criteria for Subjects in Parts 1 and 3
10. Metastatic/locally advanced solid tumor malignancy that has progressed on, is refractory to, or for which there is no standard of care therapy.
11. For subjects with cutaneous/subcutaneous lesions, subjects must have more than one measurable target lesion, at baseline, with a minimum of one lesion that meets protocol specified criteria.
12. For subjects with deep-seated lesions, subjects must have more than one measurable target lesion at baseline (RECIST v1.1), with a minimum of one deep-seated lesion suitable for image-guided injection and that meets protocol specified criteria.

    Additional Inclusion Criteria for Subjects in Part 2 (Closed to Enrollment as of Protocol Amendment 6)
13. Clinical diagnosis of CTCL, including documentation of a skin biopsy with histological findings consistent with CTCL or unconfirmed diagnosis of CTCL with confirmation biopsy at screening.
14. Stage IB, IIA, or IIB disease: T1, T2 or T3 (patches, plaques or tumors) with measurable lesions.
15. Previous treatment with at least one standard therapy used to treat the stage of disease at study entry; Stage IB, IIA or IIB CTCL.
16. Measurable skin disease with at least 2 lesions amenable to response assessment.
17. At least one lesion must be amenable to injection, ie, ≥ 1.5 cm in the longest diameter.

Exclusion Criteria:

Any of the following would exclude the subject from participation in the study:

1. Subjects who have received prior immunotherapy [(including but not limited to CTLA-4, oncolytic virus, oncolytic peptide-all require 100 day washout), programmed death ligand (PDL)-1, or programmed cell death 1 antagonists-both require 14 day washout)] are NOT permitted to enroll, with protocol exceptions.
2. Pregnant or lactating.
3. Active bacterial, fungal, or viral infections, including chronic or active hepatitis B, chronic or active hepatitis C, or active hepatitis A. Prior documented infections must have resolved.
4. Active or prior documented autoimmune or inflammatory disorders, with exceptions per protocol. Includes known allergy to sesame oil and/or nuts.
5. Immune-deficiency states - myelodysplastic disorders, marrow failures, human immunodeficiency virus (HIV) infection, history of solid organ transplant or bone marrow allograft, or recent pregnancy.
6. Requires continuous (daily) anticoagulation or antiplatelet therapy (including anti aggregants), acetylsalicylic acid (ASA) or nonsteroidal anti-inflammatory drugs (NSAIDs).
7. History of coagulopathy resulting in uncontrolled bleeding or other bleeding disorders.
8. Rapidly progressing disease per protocol.
9. Untreated or uncontrolled central nervous system (CNS) involvement.
10. Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment; with exceptions per protocol.
11. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v4.03 Grade 0 or 1, with exception of alopecia, vitiligo.
12. Uncontrolled concurrent illness.
13. Cardiac exclusions: New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled hypertension, acute coronary syndrome within 6 months, clinical important cardiac arrhythmia, mean QTC interval corrected for heart rate >500ms.
14. Major surgery within 4 weeks prior to study entry or still recovering from prior surgery.
15. Receipt of live, attenuated vaccine within 28 days prior to study entry.
16. Receipt of any systemic anticancer therapy not mentioned above within the last 2 weeks or 5 half-lives.
17. Cognitive disorder such that informed consent cannot be obtained directly from the subject
18. Subjects who have previously participated in this study and received MEDI9197, or concurrent enrollment in another clinical study involving an investigational treatment.
19. Subjects who have received prior TLR agonists, both systemic and topical.
20. Patients who have received prior therapeutic radiation within 28 days of dosing. All toxicities from prior radiotherapy must have resolved to ≤ Grade 1 or baseline prior to dosing.
21. Body weight < 35 kg
22. Subjects enrolling in Part 3 (ie, receiving durvalumab) must not have a history of interstitial lung disease or pneumonitis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by assessment of dose limiting toxicities and the maximum tolerated dose or maximal assessed dose per protocol of MEDI9197 when administered by intratumoral injection to subjects with solid tumor cancers | From time of informed consent through 4 weeks after last dose of investigational product
  The primary endpoint will be the number (%) of subjects with dose-limiting toxicities, adverse and serious adverse events and other safety parameters.
Safety and tolerability as determined by assessment of dose limiting toxicities and the maximum tolerated dose or maximal assessed dose per protocol of MEDI9197 when administered by intratumoral injection to subjects with CTCL | From time of informed consent through 6 months after last dose of investigational product
  The primary endpoint will be the number (%) of subjects with dose-limiting toxicities, adverse and serious adverse events and other safety parameters.
Safety & tolerability as determined by dose limiting toxicities and maximum tolerated or assessed dose of MEDI9197 administered by IT injection in combo with durvalumab and durvalumab plus palliative radiation to subjects with solid tumor cancers. | From time of informed consent through 90 days after last dose of investigational product
  The primary endpoint will be the number (%) of subjects with dose-limiting toxicities, adverse and serious adverse events and other safety parameters.

SECONDARY OUTCOMES:
The maximum concentration of MEDI9197 after the first injection | Pre-dose to 24 hours post first dose
The apparent terminal half-life of MEDI9197 | Pre-dose to 24 hours post first dose
Percent change from baseline in cluster of differentiation 8 tumor infiltrating lymphocytes in tumor tissue | Baseline to Day 50
Percent change from baseline in serum inflammatory cytokine levels | Pre-dose to end of study, up to 24 months
Percent change from baseline in tumor measurements | Pre-dose to disease progression, up to 12 months
Objective response rate | Pre-dose to end of study, up to 24 months
Duration of response | Pre-dose to end of study, up to 24 months
Percent change from baseline in CAILDS for subjects with CTCL | Pre-dose to disease progression, up to 12 months
Percent change from baseline in mSWAT scored for subjects with CTCL | Pre-dose to disease progression, up to 12 months
Percent change from baseline in Investigator Global Assessment (IGA) for subjects with CTCL | Pre-dose to disease progression, up to 12 months
Percent change from baseline in Subject Global Assessment (SGA) for subjects with CTCL | Pre-dose to disease progression, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (10):
- United States (8):
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
- Research Site, Toronto, Ontario, Canada
- Research Site, Villejuif, France

REFERENCES:
- [Derived] Siu L, Brody J, Gupta S, Marabelle A, Jimeno A, Munster P, Grilley-Olson J, Rook AH, Hollebecque A, Wong RKS, Welsh JW, Wu Y, Morehouse C, Hamid O, Walcott F, Cooper ZA, Kumar R, Ferte C, Hong DS. Safety and clinical activity of intratumoral MEDI9197 alone and in combination with durvalumab and/or palliative radiation therapy in patients with advanced solid tumors. J Immunother Cancer. 2020 Oct;8(2):e001095. doi: 10.1136/jitc-2020-001095. PMID 33037117